CLINICAL TRIAL: NCT00003151
Title: A Phase II Clinical Trial of Anti-Helicobacter Pylori Treatment in Endoscopically Diagnosed Low-Grade Localized Gastric Lymphoma
Brief Title: Antibiotic Therapy in Treating Patients With Low Grade Gastric Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-20961; EORTC-20961; CRC-EORTC-20961; HOVON-33
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — bismuth tripotassium dicitrate; Amoxicillin; Clarithromycin; Metronidazole; Omeprazole; Tetracycline

INTERVENTIONS:
Dietary Supplement: bismuth subcitrate
Drug: amoxicillin
Drug: clarithromycin
Drug: metronidazole hydrochloride
Drug: omeprazole
Drug: tetracycline hydrochloride

SUMMARY:
RATIONALE: Antibiotics may stop the growth of Helicobacter pylori which may be associated with gastric lymphoma.

PURPOSE: Phase II trial to study the effectiveness of antibiotic therapy in treating patients with low grade gastric lymphoma that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate of eradication of Helicobacter pylori using omeprazole, colloidal bismuth subcitrate, tetracycline, and metronidazole in patients with low grade gastric lymphoma. II. Determine the macroscopic/endoscopic and microscopic healing/remission rate after eradication of Helicobacter pylori in this patient population. III. Determine the natural history of low grade gastric lymphoma after eradication of Helicobacter pylori.

OUTLINE: This is a nonrandomized, open label, multicenter study. Patients receive oral omeprazole bid on days 1-10, oral bismuth subcitrate and oral tetracycline qid on days 4-10, and oral metronidazole tid on days 4-10. Patients are evaluated at 8 weeks. Patients who experience complete remission and are H. pylori negative proceed to follow up. Patients with complete remission or no change but who are H. pylori positive proceed to a second course of therapy with the previous schedule or with omeprazole bid, amoxicillin qid, and clarithromycin tid for 14 days. Patients who experience no change but are H. pylori negative are followed at 6 and 9 months and restaged. Patients are followed at 6, 9, 12, 18, and 24 months, then annually thereafter.

PROJECTED ACCRUAL: Approximately 60-96 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, previously untreated, low grade gastric lymphoma Clinical stage I and II1 No bulky disease No high grade component (grade 5 and 4, if monoclonality proven, allowed) Documented presence/absence of H. pylori infection Measurable and/or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or lactating Fertile patients must use effective contraception No prior or concurrent malignancies unless: At least 1 year remission Low risk or recurrence No prior gastric malignancy No nonmalignant disease causing poor medical risk No allergy to omeprazole

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the abdomen Surgery: No prior gastric surgery except simple closure of perforated ulcer with or without wedge excision of the ulcer Other: No prior therapy for gastric lymphoma At least 30 days since experimental therapy No other concurrent experimental therapy At least 30 days since antibiotics with activity against H. pylori

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 1997-09; Primary Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P. Carde, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; John W. Sweetenham, MD, Study Chair — University of Colorado, Denver
Locations (22):
- United Kingdom (22):
  - Royal United Hospital, Bath, England
  - University Birmingham N.H.S. Trust, Birmingham, England
  - Royal Free Hospital, Hampstead, London, England
  - St. James's Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Free Hospital School of Medicine, London, England
  - Guy's, King's and St. Thomas' Hospitals Trust, London, England
  - Royal Marsden NHS Trust, London, England
  - Hammersmith Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Charing Cross Hospital, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Royal South Hants Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Infirmary, Glasgow, Scotland